CLINICAL TRIAL: NCT03756077
Title: A Prospective Study of the Value of Hybrid PET/MR and PET/CT in Prostate Cancer
Brief Title: A Study of the Value of Hybrid PET/MR and PET/CT in Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaoli Lan, Director of the Department of nuclear medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: XLan
Record Dates: First submitted 2018-11-25; First posted 2018-11-28 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Prostate Cancer; PET/MR; PET/CT
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary diagnosis and staging: Patients suspected of or diagnosed with prostate cancer who want a differential diagnosis and staging by 68Ga-PSMA-11 and/or 18F-FDG PET/MR, PET/CT before treatment
  Interventions: Diagnostic Test: 68Ga-PSMA-11 and/or 18F-FDG PET/MR, PET/CT
- Evaluation of recurrence: Patients with a history of prostate cancer and elevated PSA level after treatment, who need to determining whether or not there are recurrences/metastatic lesions and its locations by 68Ga-PSMA-11 and/or 18F-FDG PET/MR, PET/CT
  Interventions: Diagnostic Test: 68Ga-PSMA-11 and/or 18F-FDG PET/MR, PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-PSMA-11 and/or 18F-FDG PET/MR, PET/CT — 0.05-0.06 mCi per kilogram bodyweight of 68Ga-PSMA, 0.1-0.15 mCi per kilogram bodyweight of 18F-FDG will be injected intravenously prior to imaging

SUMMARY:
According to the latest data from the China National Cancer Center, prostate cancer has become the most common tumor in the urinary system since 2008. However, conventional imaging techniques including transrectal ultrasound , computed tomography and bone scintigraphy are not sensitive or specific. About 40% of resectable lesions cannot be detected by these techniques. Positron Emission Tomography (PET) provides a valuable tool for the diagnosis and staging of prostate cancer. Recently, prostate-specific membrane antigen (PSMA) as a new novel positron tracer has shown to be effective to detect primary lesions, recurrent and metastatic lesions of prostate cancer. In this prospective study, the investigators will use the most advanced imaging equipments, integrated PET/MR, and PET/CT with prostate cancer-specific imaging agent 68Ga-PSMA and conventional imaging agent [F-18]fluorodeoxyglucose to image patients with or suspected of prostate cancer, the aim is to explore the value of hybrid PET/MR and PET/CT in prostate cancer.

DETAILED DESCRIPTION:
According to the latest data from the China National Cancer Center, prostate cancer has become the most common tumor in the urinary system since 2008. However, conventional imaging techniques including transrectal ultrasound , computed tomography and bone scintigraphy are not sensitive or specific. About 40% of resectable lesions cannot be detected by these techniques. Positron Emission Tomography (PET) provides a valuable tool for the diagnosis and staging of prostate cancer. Recently, prostate-specific membrane antigen (PSMA) as a new novel positron tracer has shown to be effective to detect primary lesions, recurrence and metastatic lesions of prostate cancer. In this prospective study, the investigators will use the most advanced imaging equipment, integrated PET/MR, and PET/CT with prostate cancer-specific imaging agent 68Ga-PSMA and conventional imaging agent [F-18]fluorodeoxyglucose to image patients. For patients suspected of or diagnosed with prostate cancer, the investigators aim to evaluate the roles of integrated PET/MR and PET/CT in differential diagnosis, detecting primary and metastatic lesions, guilding biopsy, staging and determining treatment plan prior to treatment; for the patients with a history of prostate cancer, the aim is to evaluate the value of integrated PET/MR and PET/CT for treatment response assessment, detection of recurrences and metastatic lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected of or diagnosed with prostate cancer

Exclusion Criteria:

* Acute systemic diseases and electrolyte disorders
* Patients with known malignancy in other organs
* Patients with severe claustrophobia or unstable vital sigh
* Other serious comorbidities evaluated by primary investigator

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Central China
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-04-26 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of 68Ga- PSMA, 18F-FDG PET/MR, PET/CT for initial diagnosis and staging | up to 2 years
  For patient without any treatment, Initial diagnosis and staging results of 68Ga- PSMA, 18F-FDG PET/MR, PET/CT will be compared to pathology, clinical and follow-up result. Evaluation of the concordance between 68Ga-PSMA PET/MR and PET/CT, the differences between 68Ga-PSMA and 18F-FDG.

SECONDARY OUTCOMES:
Sensitivity and specificity of 68Ga- PSMA, 18F-FDG PET/MR, PET/CT for recurrence detection | up to 2 years
  For patient with a history of prostate cancer, results of 68Ga- PSMA, 18F-FDG PET/MR, PET/CT will be compared to pathology, clinical and follow-up result. Evaluation of the concordance between 68Ga-PSMA PET/MR and PET/CT, the differences between 68Ga-PSMA and 18F-FDG.
Sensitivity of 68Ga-PSMA PET/MR, PET/CT for different PSA levels, different lesion sites | up to 2 years
  For patient with a history of prostate cancer and suspected of recurrence, evaluate Sensitivity and specificity of 68Ga- PSMA, 18F-FDG PET/MR, PET/CT for different PSA levels, different lesion sites

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Lan, MD, PhD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Xiaoli Lan, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Qin C, Gai Y, Liu Q, Ruan W, Liu F, Hu F, Zhang X, Lan X. Optimized Application of 68Ga-Prostate-Specific Membrane Antigen-617 Whole-Body PET/CT and Pelvic PET/MR in Prostate Cancer Initial Diagnosis and Staging. Front Med (Lausanne). 2021 May 13;8:657619. doi: 10.3389/fmed.2021.657619. eCollection 2021. PMID 34055836